CLINICAL TRIAL: NCT07226089
Title: Multicenter Interventional Study: Somatrogon Impact on Outcomes in Naive Small for Gestational Age or Idiopathic Short Stature Pediatric Patients Compared With Daily Growth Hormone
Brief Title: Comparison of Weekly Somatrogon to Daily Genotropin in Children Born Small for Gestational Age or With Idiopathic Short Stature.
Acronym: MISSION
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0081-24-RMC
Record Dates: First submitted 2025-11-06; First posted 2025-11-10 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: ISS; SGA
Keywords: Growth hormone; Somatrogon
MeSH Terms: interventions — somatrogon; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Somatrogon (Experimental): Somatrogon will be administered subcutaneously (s.c) once weekly using a multi dose disposable prefilled pen for single patient use intended for SC self injection.
  Interventions: Drug: Somatrogon
- Genotropin (Active Comparator): Genotropin will be administrated subcutaneously (s.c) daily using Genotropin Pen growth hormone delivery devices or Genotropin two chamber cartridges (will be supplied in their primary commercial packaging)
  Interventions: Drug: Genotropin

INTERVENTIONS:
Drug: Somatrogon — Once weekly Growth Hormone
  Other Names: NGENLA 60mg SSOL 1x1.2mL PFP US
  Arms: Somatrogon
Drug: Genotropin — Daily Growth Hormone
  Other Names: Genotropin PEN 12 1x U2 US
  Arms: Genotropin

SUMMARY:
This study is a randomized, open-label, active controlled, parallel group study comparing the efficacy and safety of once weekly Somatrogon to daily Growth Hormone (Genotropin) in pre-pubertal children with short stature either born Small for Gestational Age (SGA) or with Idiopathic Short Stature (ISS). The planned study duration is 12 months with a screening period of up to 30 days. The study will consist of two groups: 140 children with SGA who are naïve to GH treatment will be randomized 1:1 to receive either Somatrogon or Genotropin for 12 months. A second group will include 114 children with ISS who are naïve to GH treatment who will be randomized 1:1 to receive either Somatrogon or Genotropin for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of SGA or ISS. SGA, defined as born with a birth weight and/or length <-2 SDS below the mean for gestational age. ISS, defined as height < -2 SDS for age and gender without evidence of GHD
2. Females aged ≥3 years and <9 years. Males aged ≥3 years and <11 years
3. Pre-pubertal- Tanner stage 1 for breasts and testes.
4. A bone age of not more than chronological age recorded in previous 8 weeks.
5. Current height < -2 SDS for age and gender.
6. Participants using hormonal replacement therapy(s) must be on an optimized and stable treatment regimen (hormone levels within normal ranges on screening) for at least three months prior to screening
7. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. History of cancer, radiation therapy or chemotherapy.
2. History of GHD.
3. Children who are small due to malnutrition, defined as a Z score of weight for height and/or BMI below -2 for age, according to national standards.
4. History of HIV-positive, acquired immune deficiency syndrome (AIDS), hepatitis B, hepatitis C, or tuberculosis.
5. Microcephaly (Head Circumference < -2 SDS)
6. Any chronic disease or diagnosis, likely to affect growth, including but not limited to gastrointestinal disorder, celiac disease, untreated thyroid disease, diabetes mellitus and metabolic disorders.
7. Known or suspected skeletal dysplasias
8. Known or suspected chromosomal abnormalities
9. IGF-1 >2 SDS
10. Any disorder or condition which, in the opinion of the investigator, might jeopardize participant's safety or compliance with the protocol
11. Prior exposure to growth promoting therapy
12. Current use of any prohibited concomitant medication(s): Any rhGH or growth-promoting therapy, Any therapy that affects appetite or weight, Psychiatric medications associated with weight changes and/or diabetes, excluding medications used to treat ADHD, Any androgen or estrogen therapy including over the counter supplements, Systemic corticosteroids (inhaled or oral) exceeding the doses: Inhaled: > 400 μg/day of inhaled budesonide or equivalent. Oral: > 8 mg/m2/day of oral hydrocortisone or equivalent.
13. Previous administration with an investigational drug within 90 days.
14. Fasting blood glucose >126 mg/dL
15. Renal impairment
16. Hepatic dysfunction.
17. Pregnancy
18. Known hypersensitivity to the components of the study intervention

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 254 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Annual Height Velocity | • Annualized HV after 12 months of treatment
  Annual Height Velocity in cm. Annual Height Velocity at 12 months is based on the difference between the heights at 12 months and baseline.

SECONDARY OUTCOMES:
Height Velocity over time | HV over 3, 6 and 9 months
height SDS | 3, 6, 9 and 12 months
  Changes in height Standard Deviation Score (SDS)
Bone maturation | at screening and after 12 months
  Annual change in bone age measurements as per Gruelich-Pyle method
Insulin-like Growth Factor-1 (IGF-1) | Screening and after 3, 6, 9 and 12 months
  Via central lab analysis
Insulin-like Growth Factor-1 (IGF-1) Standard Deviation Score (SDS) | Baseline and at 12 months
  Via central lab analysis
change in health-related quality of life | baseline and after 12 months
  Assessed by QoLISSY questionnaire

OTHER OUTCOMES:
IGFBP-3 | At baseline and after 12 months
  Via central lab
Frequency of abnormal lab results in the Somatrogon arm | At screening, baseline and after 1, 3, 6 ,9 and 12 months
SAE's in the Somatrogon arm | At screening, baseline and after 1, 3, 6 ,9 and 12 months
AE's in the Somatrogon arm | At screening, baseline and after 1, 3, 6 ,9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Professor, Study Director — Schneider Children's Medical Center
Locations (6):
- Israel (6):
  - Schneider Children Medical Center- the institute of Endocrinology and Diabetes, Petah Tikva, Israel
  - Shaare Zedek Medical Center, Jerusalem, Israe
  - Soroka hospital, Bear Sheva
  - Sheba Medical Center, Ramat Gan
  - Assaf Harofe Medical Center, Rishon LeZiyyon
  - Dana-Duek children's hospital, Tel Aviv

IPD SHARING:
Plan to Share IPD: No
We would only share patient data with regulatory agencies that require the information.